CLINICAL TRIAL: NCT03348904
Title: A Phase 3, Randomized, Global Trial of Nivolumab and Epacadostat With Platinum Doublet Chemotherapy Versus Platinum Doublet Chemotherapy in First-line Treatment of Stage IV or Recurrent Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Nivolumab and Epacadostat With Platinum Doublet Chemotherapy Versus Platinum Doublet Chemotherapy in Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study halted prematurely and will not resume; participants are no longer being examined or receiving intervention.
Sponsor: Incyte Corporation (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA2099NC/ECHO-309
Record Dates: First submitted 2017-11-16; First posted 2017-11-21 (Actual); Results first posted 2019-06-13 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Lung Cancer
Keywords: Non-small cell lung cancer; programmed cell death protein 1 (PD-1) antibody; indoleamine 2,3-dioxygenase (IDO) inhibitor
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — Nivolumab; epacadostat; Carboplatin; Cisplatin; Gemcitabine; Paclitaxel; Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): Nivolumab plus epacadostat in combination with platinum doublet
  Interventions: Drug: Nivolumab; Drug: Epacadostat; Drug: Carboplatin; Drug: Cisplatin; Drug: Gemcitabine; Drug: Paclitaxel; Drug: Pemetrexed
- Arm B (Active Comparator): Platinum doublet chemotherapy
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Gemcitabine; Drug: Paclitaxel; Drug: Pemetrexed
- Arm C (Experimental): Nivolumab plus placebo in combination with platinum doublet chemotherapy.
  Interventions: Drug: Nivolumab; Drug: Placebo; Drug: Carboplatin; Drug: Cisplatin; Drug: Gemcitabine; Drug: Paclitaxel; Drug: Pemetrexed

INTERVENTIONS:
Drug: Nivolumab — Nivolumab administered intravenously at the protocol-defined dose every 3 weeks.
  Other Names: BMS-936558
  Arms: Arm A; Arm C
Drug: Epacadostat — Epacadostat administered orally at the protocol-defined dose twice daily.
  Other Names: INCB024360
  Arms: Arm A
Drug: Placebo — Matching placebo for epacadostat administered orally twice daily.
  Arms: Arm C
Drug: Carboplatin — Carboplatin administered intravenously at the protocol-defined dose every 3 weeks for up to 4 cycles.
Drug: Cisplatin — Cisplatin administered intravenously at the protocol-defined dose every 3 weeks for up to 4 cycles.
Drug: Gemcitabine — Gemcitabine administered intravenously at the protocol-defined dose every 3 weeks for up to 4 cycles.
Drug: Paclitaxel — Paclitaxel administered intravenously at the protocol-defined dose every 3 weeks for up to 4 cycles.
Drug: Pemetrexed — Pemetrexed administered intravenously at the protocol-defined dose every 3 weeks for up to 4 cycles. Optional continuation maintenance every 3 weeks, if eligible.

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of the combination of nivolumab plus epacadostat in combination with platinum chemotherapy compared with platinum chemotherapy alone, in participants with treatment-naïve Stage 4 or recurrent non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage IV or recurrent NSCLC of squamous or non-squamous histology that is not amenable to therapy with curative intent (surgery or radiation therapy with or without chemotherapy).
* No prior treatment with systemic anti-cancer therapy for Stage IV disease.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to1.
* Measurable disease by computed tomography or magnetic resonance imaging per RECIST v1.1.
* Documentation of program death ligand-1 (PD-L1) status of 0 to 49% by IHC performed by the central laboratory prior to randomization.
* Other protocol inclusion criteria may apply

Exclusion Criteria:

* Known epidermal growth factor receptor (EGFR) mutations sensitive to available targeted inhibitor therapy.
* Known ALK or ROS1 rearrangements sensitive to available targeted inhibitor therapy.
* Untreated central nervous system (CNS) metastases.
* Unevaluable PD-L1 status or PD-L1 status of ≥ 50% by IHC performed by a central laboratory.
* Carcinomatous meningitis.
* Active, known or suspected autoimmune disease.
* Prior treatment with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, IDO1 targeted agent, or any other antibody or drug targeting T cell co-stimulation or checkpoint pathways.
* History of allergy or hypersensitivity to platinum-containing compounds or study drug components.
* Physical and laboratory test findings outside the protocol-defined range.
* Other protocol exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-12-27 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2018-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sridhar K. Rabindran, PhD, Study Director — Bristol-Myers Squibb Research and Development
Locations (2):
- United States (2):
  - Pacific Cancer Medical Center, Inc, Anaheim, California
  - Cancer Center of Kansas, Wichita, Kansas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 630 participants were planned to be randomized. Prior to the termination of the study, 2 participants were randomized to the Platinum Doublet Chemotherapy arm (Arm B) and treated.
Groups:
- Nivolumab + Epacadostat/Platinum Doublet Chemotherapy: Nivolumab + Epacadostat/Platinum Doublet Chemotherapy included the following:
  Nivolumab was administered intravenously at the protocol-defined dose every 3 weeks. Epacadostat was administered orally at the protocol-defined dose twice daily. Carboplatin was administered intravenously at the protocol-defined dose every 3 weeks for up to 4 cycles. Cisplatin was administered intravenously at the protocol-defined dose every 3 weeks up to 4 cycles. Gemcitabine was administered intravenously at the protocol-defined dose every 3 weeks up to 4 cycles. Paclitaxel was administered intravenously at the protocol-defined dose every 3 weeks up to 4 cycles. Pemetrexed was administered intravenously at the protocol-defined dose every 3 weeks up to 4 cycles.
  Optional continuation maintenance was available every 3 weeks, if eligible.
- Platinum Doublet Chemotherapy: Platinum Doublet Chemotherapy included the following:
  Carboplatin was administered intravenously at the protocol-defined dose every 3 weeks up to 4 cycles. Cisplatin was administered intravenously at the protocol-defined dose every 3 weeks up to 4 cycles. Gemcitabine was administered intravenously at the protocol-defined dose every 3 weeks up to 4 cycles. Paclitaxel was administered intravenously at the protocol-defined dose every 3 weeks up to 4 cycles. Pemetrexed was administered intravenously at the protocol-defined dose every 3 weeks up to 4 cycles.
  Optional continuation maintenance was available every 3 weeks, if eligible.
- Nivolumab + Placebo Combination/Platinum Doublet Chemotherapy: Nivolumab plus placebo in combination with platinum doublet chemotherapy included:
  Nivolumab was administered intravenously at the protocol-defined dose every 3 weeks. : Matching placebo for epacadostat was administered orally twice daily. Carboplatin was administered intravenously at the protocol-defined dose every 3 weeks up to 4 cycles. Cisplatin was administered intravenously at the protocol-defined dose every 3 weeks up to 4 cycles. Gemcitabine was administered intravenously at the protocol-defined dose every 3 weeks up to 4 cycles. Paclitaxel was administered intravenously at the protocol-defined dose every 3 weeks up to 4 cycles. Pemetrexed was administered intravenously at the protocol-defined dose every 3 weeks up to 4 cycles.
  Optional continuation maintenance was available every 3 weeks, if eligible.
Period: Overall Study
Arm/Group | Nivolumab + Epacadostat/Platinum Doublet Chemotherapy | Platinum Doublet Chemotherapy | Nivolumab + Placebo Combination/Platinum Doublet Chemotherapy
Started | 0 | 2 | 0
Completed | 0 | 1 | 0
Not Completed | 0 | 1 | 0
Not completed — Administrative reason by the sponsor | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab + Epacadostat/Platinum Doublet Chemotherapy | Platinum Doublet Chemotherapy | Nivolumab + Placebo Combination/Platinum Doublet Chemotherapy | Total
Number analyzed (Participants) | 0 | 2 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 2 | 0 | 2
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 0 | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White or Caucasian | 0 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) of Nivolumab Plus Epacadostat in Combination With Chemotherapy (Arm A) Compared to Chemotherapy (Arm B)
Description: Defined as the time from randomization to the date of death from any cause.
Time Frame: Approximately 38 months
Population: All randomized participants; Arm A did not enroll any participants in the study and as a result no comparisons were performed and since the study was terminated early no efficacy analyses were conducted.
Arm/Group | Nivolumab + Epacadostat/Platinum Doublet Chemotherapy | Platinum Doublet Chemotherapy
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Progression-free Survival (PFS) of Nivolumab Plus Epacadostat in Combination With Chemotherapy (Arm A) Compared to Chemotherapy (Arm B)
Description: Defined as the time between the date of randomization and the first date of documented progression assessed by blinded independent central review, or death due to any cause, whichever occurs first.
Time Frame: Approximately 25 months
Population: as for outcome 1
Arm/Group | Nivolumab + Epacadostat/Platinum Doublet Chemotherapy | Platinum Doublet Chemotherapy
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Objective Response Rate (ORR) of Nivolumab Plus Epacadostat in Combination With Chemotherapy (Arm A) Compared to Chemotherapy (Arm B)
Description: Defined as the proportion of participants who achieve a confirmed best response of complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) criteria as assessed by blinded independent central review.
Time Frame: Approximately 25 months
Population: as for outcome 1
Arm/Group | Nivolumab + Epacadostat/Platinum Doublet Chemotherapy | Platinum Doublet Chemotherapy
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Duration of Response (DOR) of Nivolumab Plus Epacadostat in Combination With Chemotherapy (Arm A) Compared to Chemotherapy (Arm B)
Description: Defined as the time between the date of first confirmed response and the date of the first documented tumor progression (per RECIST v1.1) assessed by blinded independent central review or death due to any cause, whichever occurs first.
Time Frame: Approximately 25 months
Population: as for outcome 1
Arm/Group | Nivolumab + Epacadostat/Platinum Doublet Chemotherapy | Platinum Doublet Chemotherapy
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Estimate of OS of Nivolumab and Placebo in Combination With Chemotherapy (Arm C)
Description: Defined as the time from randomization to the date of death from any cause.
Time Frame: Approximately 38 months
Population: All randomized participants; Arm C did not enroll any participants in the study and as a result no analyses were performed and since the study was terminated early no efficacy analyses were conducted.
Arm/Group | Nivolumab + Placebo Combination/Platinum Doublet Chemotherapy
Number analyzed (Participants) | 0

6. Secondary Outcome: Estimate of PFS of Nivolumab and Placebo in Combination With Chemotherapy (Arm C)
Description: Defined as the time between the date of randomization and the first date of documented progression assessed by blinded independent central review or death due to any cause, whichever occurs first.
Time Frame: Approximately 25 months
Population: as for outcome 5
Arm/Group | Nivolumab + Placebo Combination/Platinum Doublet Chemotherapy
Number analyzed (Participants) | 0

7. Secondary Outcome: Estimate of ORR of Nivolumab and Placebo in Combination With Chemotherapy (Arm C)
Description: Defined as the proportion of participants who achieve a confirmed best response of CR or PR per RECIST v1.1 criteria as assessed by blinded independent central review.
Time Frame: Approximately 25 months
Population: as for outcome 5
Arm/Group | Nivolumab + Placebo Combination/Platinum Doublet Chemotherapy
Number analyzed (Participants) | 0

8. Secondary Outcome: Estimate of DOR of Nivolumab and Placebo in Combination With Chemotherapy (Arm C)
Description: as for outcome 4
Time Frame: Approximately 25 months
Population: as for outcome 5
Arm/Group | Nivolumab + Placebo Combination/Platinum Doublet Chemotherapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From the initiation of study treatment until 30 days after last dose of study treatment or up to study termination date 22May2018.
Description: All treated participants.
Arm/Group | Nivolumab + Epacadostat/Platinum Doublet Chemotherapy | Platinum Doublet Chemotherapy | Nivolumab + Placebo Combination/Platinum Doublet Chemotherapy
All-Cause Mortality (participants affected / at risk) | 0/0 | 1/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 1/2 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 2/2 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + Epacadostat/Platinum Doublet Chemotherapy (N=0) | Platinum Doublet Chemotherapy (N=2) | Nivolumab + Placebo Combination/Platinum Doublet Chemotherapy (N=0)
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + Epacadostat/Platinum Doublet Chemotherapy (N=0) | Platinum Doublet Chemotherapy (N=2) | Nivolumab + Placebo Combination/Platinum Doublet Chemotherapy (N=0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (1):
  • Study Protocol (2017-10-23): https://cdn.clinicaltrials.gov/large-docs/04/NCT03348904/Prot_000.pdf